CLINICAL TRIAL: NCT02517775
Title: Intake and Time-dependent Effects of Cranberry (Poly)Phenol Consumption in Vascular Function in Healthy Individuals
Brief Title: Effects of Cranberry Consumption in Vascular Function in Healthy Individuals
Acronym: Cranberry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: The Cranberry Institute (Other)
Responsible Party: Principal Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Division of Cardiology, Pulmonary Diseases, Vascular Medicine, Heinrich-Heine University, Duesseldorf
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 14-012
Record Dates: First submitted 2015-07-08; First posted 2015-08-07 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Healthy Men
Keywords: polyphenols; vascular function; endothelial function; cranberry; healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cranberry 320 (Active Comparator): Dietary Supplement: Cranberry beverage with 320 mg of (poly)phenols Acute intake of 500 mL (1x daily)
  Interventions: Dietary Supplement: Cranberry 320
- Cranberry 640 (Active Comparator): Dietary Supplement: Cranberry beverage with 640 mg of (poly)phenols Acute intake of 500 mL (1x daily)
  Interventions: Dietary Supplement: Cranberry 640
- Cranberry 960 (Active Comparator): Dietary Supplement: Cranberry beverage with 960 mg of (poly)phenols Acute intake of 500 mL (1x daily)
  Interventions: Dietary Supplement: Cranberry 960
- Cranberry 1280 (Active Comparator): Dietary Supplement: Cranberry beverage with 1280 mg of (poly)phenols Acute intake of 500 mL (1x daily)
  Interventions: Dietary Supplement: Cranberry 1280
- Cranberry 1600 (Active Comparator): Dietary Supplement: Cranberry beverage with 1600 mg of (poly)phenols Acute intake of 500 mL (1x daily)
  Interventions: Dietary Supplement: Cranberry 1600
- Cranberry deprived supplement (Placebo Comparator): Placebo comparator: Cranberry deprived supplement Acute intake of 500 mL (1x daily)
  Interventions: Dietary Supplement: Cranberry deprived supplement

INTERVENTIONS:
Dietary Supplement: Cranberry 320 — Dietary Supplement: Cranberry beverage with 320 mg of (poly)phenols Acute intake of 500 mL (1x daily)
  Arms: Cranberry 320
Dietary Supplement: Cranberry 640 — Dietary Supplement: Cranberry beverage with 640 mg of (poly)phenols Acute intake of 500 mL (1x daily)
  Arms: Cranberry 640
Dietary Supplement: Cranberry 960 — Dietary Supplement: Cranberry beverage with 960 mg of (poly)phenols Acute intake of 500 mL (1x daily)
  Arms: Cranberry 960
Dietary Supplement: Cranberry 1280 — Dietary Supplement: Cranberry beverage with 1280 mg of (poly)phenols Acute intake of 500 mL (1x daily)
  Arms: Cranberry 1280
Dietary Supplement: Cranberry 1600 — Dietary Supplement: Cranberry beverage with 1600 mg of (poly)phenols Acute intake of 500 mL (1x daily)
  Arms: Cranberry 1600
Dietary Supplement: Cranberry deprived supplement — Cranberry deprived supplement Acute intake of 500 mL (1x daily)
  Arms: Cranberry deprived supplement

SUMMARY:
Accumulating evidence from epidemiological and human intervention studies indicates that the cardiovascular health benefits of diets rich in fruits and vegetables are (in part) related to their (poly)phenol content. Cranberries are rich in (poly)phenols compounds, in particular anthocyanins, but also phenolic acids. At present, a small number of randomized controlled trials investigating the effects of berry (poly)phenols on validated surrogate markers of cardiovascular disease risk has shown promising results. However, to date, very few human studies have specifically investigated the effects of cranberry (poly)phenols on cardiovascular function in healthy subjects. To our knowledge, no study has investigated the time and intake-dependent effect of cranberry consumption on vascular function in healthy subjects. This information is necessary for the planning of long-term studies aiming to assess the potential beneficial effects of cranberries, using optimal amounts at optimal time points. Therefore, this study aims to investigate the potential role of cranberry (poly)phenols in the modulation of vascular function by monitoring changes in vascular function together with the major (poly)phenol derivatives/metabolites in plasma and urine.

ELIGIBILITY:
Inclusion Criteria:

* healthy male subjects without clinical signs or symptoms of cardiovascular disease

Exclusion Criteria:

* cardiovascular disease
* acute inflammation
* cardiac arrhythmia
* renal failure
* heart failure (NYHA II-IV)
* diabetes mellitus
* C-reactive protein > 05 mg/dL
* malignant disease
* cranberry allergy/intolerance
* hypotension (≤100 / 60 mm Hg)

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Endothelial function | Baseline, on week 1, 2, 3, 4 and 5 postconsumption
  measured by Flow mediated dilation at 1, 2, 4, 6 and 8 hours after intake

SECONDARY OUTCOMES:
pulse wave velocity | Baseline, on week 1, 2, 3, 4 and 5 postconsumption
  measured by SphygmoCor at 0, 1, 2, 4, 6 and 8 hours after intake
Central blood pressure | Baseline, on week 1, 2, 3, 4 and 5 postconsumption
  measured by SphygmoCor at 0, 1.5, 4, 6 and 8 hours after intake
Peripheral blood pressure | Baseline, on week 1, 2, 3, 4 and 5 postconsumption
  measured by automatic sphygmomanometer at 0, 1, 2, 4, 6 and 8 hours after intake
Heart Rate | Baseline, on week 1, 2, 3, 4 and 5 postconsumption
  measured by SphygmoCor 0, 1, 2, 4, 6 and 8 hours after intake

OTHER OUTCOMES:
Plasma (poly)phenol metabolites | Baseline, on week 1, 2, 3, 4 and 5 postconsumption
  measured by ultra-performance liquid chromatography quadrupole time of flight mass spectrometry (UPLC-Q-TOF MS) at 0,1, 2, 4, 6, 8 and 24 hours after intake
Urinary (poly)phenol metabolites | Baseline, on week 1, 2, 3, 4 and 5 postconsumption
  measured by ultra-performance liquid chromatography quadrupole time of flight mass spectrometry (UPLC-Q-TOF MS) at 0, 8 and 24 hours after intake

CONTACTS AND LOCATIONS:
Overall Officials: Ana Rodriguez-Mateos, PhD, Principal Investigator — Division of Cardiology, Pulmonology and Vascular Medicine; Christian Heiss, MD, Principal Investigator — Division of Cardiology, Pulmonology and Vascular Medicine
Locations (1):
- Division of Cardiology, Pulmonary Disease and Vascular Medicine, University Hospital Duesseldorf, Düsseldorf, Germany

REFERENCES:
- [Derived] Mena P, Favari C, Acharjee A, Chernbumroong S, Bresciani L, Curti C, Brighenti F, Heiss C, Rodriguez-Mateos A, Del Rio D. Metabotypes of flavan-3-ol colonic metabolites after cranberry intake: elucidation and statistical approaches. Eur J Nutr. 2022 Apr;61(3):1299-1317. doi: 10.1007/s00394-021-02692-z. Epub 2021 Nov 9. PMID 34750642